CLINICAL TRIAL: NCT03703908
Title: An Open Label, Intra-Subject Dose Escalation Study of CCX140-B in Subjects With Primary Focal Segmental Glomerulosclerosis (FSGS) and Nephrotic Syndrome
Brief Title: A Study of CCX140-B in Subjects With Primary FSGS and Nephrotic Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Program not advancing
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CL012_140; LUMINA-2 (Other: Chemocentryx)
Record Dates: First submitted 2018-07-24; First posted 2018-10-12 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Focal Segmental Glomerulosclerosis
Keywords: FSGS; Glomerulosclerosis; Proteinuria
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Proteinuria | interventions — CCX140-B

STUDY DESIGN:
Intervention Model Description: Open-Label, Intra-Subject, Dose Escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sequential (Experimental): All enrolled subjects will initially be treated with the active study medication CCX140-B at a dose of 5 mg twice daily. Dose will increase in a step-wise fashion up to 15 mg twice daily.
  Interventions: Drug: CCX140-B

INTERVENTIONS:
Drug: CCX140-B — Orally administered tablet

SUMMARY:
An Open Label, Intra-Subject Dose Escalation Study of CCX140 B in Subjects with Primary FSGS and Nephrotic Syndrome

DETAILED DESCRIPTION:
An Open Label, Intra-Subject Dose Escalation Study of CCX140 B in Subjects with Primary Focal Segmental Glomerulosclerosis (FSGS) and Nephrotic Syndrome. The aim of this study is to explore the effect of CCX140-B, a selective antagonist of C-C chemokine receptor type 2, on proteinuria in subjects with FSGS.

Study acquired by Amgen and all disclosures were done by previous sponsor ChemoCentryx.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 years and older
2. Primary FSGS based on renal biopsy findings consistent with FSGS and based on presentation of histopathology, medical history and clinical course OR subjects with genetic risk factors with presentations that are otherwise consistent with primary FSGS
3. Urinary total protein:creatinine ratio (UPCR) ≥ 3.5 g protein/g creatinine at screening

Exclusion Criteria:

1. Pregnant or nursing
2. History of organ transplantation, including renal transplantation
3. Currently on an organ transplant waiting list or there's a reasonable possibility of getting an organ transplant within 6 months of screening
4. Histological FSGS subtype of collapsing variant
5. Subjects who initiated, discontinued or changed dose of anti-CD20 monoclonal antibodies within 16 weeks (4 months) prior to screening are excluded. Subjects who initiated treatment with anti-CD20 monoclonal antibodies >16 weeks (4 months) prior to screening are permitted if deemed safe by the investigator and only if they intend to remain on continued, unchanged therapy at a dosing interval that has been documented to achieve continuous B cell depletion for the given patient.
6. Subjects who discontinued Rituximab or other anti-CD20 monoclonal antibodies >16 weeks (4 months) prior to screening without confirmed recovery of CD20+ B cell population to within normal range are excluded. Subjects who discontinued rituximab or other anti-CD20 monoclonal antibodies >16 weeks (4 months) prior to screening with confirmed recovery of CD20+ B cell population to within normal range are permitted in the study. UPCR and other urine protein assessments up to 1 year prior to screening (if available) that were performed in these patients as part of the clinical routine should be recorded in the medical history.
7. Body Mass Index (BMI) ≥ 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (5):
- United States (5):
  - Los Angeles Biomedical Research Institute, Torrance, California
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Utah Kidney Research Institute, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- CCX140-B: Drug: CCX140-B, orally administered tablet All enrolled subjects will initially be treated with the active study medication CCX140-B at a dose of 5 mg twice daily. Dose will increase in a step-wise fashion up to 15 mg twice daily.
Period: Overall Study
Arm/Group | CCX140-B
Started | 5
Completed | 2
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- CCX140-B: CCX140-B is an orally administered tablet All enrolled subjects will initially be treated with the active study medication CCX140-B at a dose of 5 mg twice daily. Dose will increase in a step-wise fashion up to 15 mg twice daily.
Arm/Group | CCX140-B
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (18.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4
  Poland | 1
Age at diagnosis of FSGS (years) [Mean (Standard Deviation); unit: years] — FSGS= Focal segmental glomerulosclerosis
  years | 35.2 (19.18)
Duration of FSGS (months) [Mean (Standard Deviation); unit: months] — Duration of Focal segmental glomerulosclerosis (FSGS) was calculated from the time of first diagnosis based on renal biopsy.
  months | 29.4 (16.32)
Baseline UPCR - morning void [Mean (Standard Deviation); unit: g protein/ g creatinine] — UPCR= Urine protein:creatinine ratio
  g protein/ g creatinine | 5.71 (1.563)
Baseline UPCR - 24-hour [Mean (Standard Deviation); unit: g protein/ g creatinine] | 4.80 (1.376)
Baseline UACR - morning void [Mean (Standard Deviation); unit: g protein/ g creatinine] — UACR= Urinary albumin:creatinine ratio
  g protein/ g creatinine | 4.12 (1.394)
Baseline UACR - 24-hour [Mean (Standard Deviation); unit: g protein/ g creatinine] | 3.24 (1.316)
Concomitant use of glucocorticoids and/or immunosuppressive medications [Count of Participants; unit: Participants]
  Yes | 4
  No | 1
Concomitant use of ACE inhibitor or ARB [Count of Participants; unit: Participants] — ACE= Angiotensin-converting enzyme, ARB= Angiotensin receptor blocker
  Participants
    Yes | 5
    No | 0
All calcineurin inhibitors combined [Count of Participants; unit: Participants] — Includes cyclosporin or tacrolimus
  Participants
    Yes | 2
    No | 3
Concomitant use of rituximab or other anti-CD20 [Count of Participants; unit: Participants]
  Yes | 0
  No | 5
Baseline eGFR (CKD-EPI Creatinine-Cystatin C) [Mean (Standard Deviation); unit: mL/min/1.73m²] — eGFR= Estimated glomerular filtration rate, CKD-EPI= Chronic Kidney Disease Epidemiology Collaboration
  mL/min/1.73m² | 50.60 (23.923)
Baseline eGFR (MDRD Creatinine) [Mean (Standard Deviation); unit: mL/min/1.73m²] — MDRD= Modification of Diet in Renal Disease
  mL/min/1.73m² | 54.40 (26.245)
Podocyte effacement [Count of Participants; unit: Participants] — Based on electron microscopy
  Participants
    <30% | 1
    ≥30% | 4
Glomeruli showing segmental lesions [Count of Participants; unit: Participants]
  ≤1 | 1
  >1 | 4

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects With a Reduction in Urine Protein to Creatinine Ratio (UPCR) of at Least 20%
Description: Number of subjects with a reduction in Urine Protein to Creatinine Ratio (UPCR) of at least 20% , i.e., ≥20%, by Week 12.
Time Frame: Baseline to week 12
Measure: Count of Participants; unit: Participants
Arm/Group | CCX140-B
Number analyzed (Participants) | 5
Participants | 2

2. Secondary Outcome: Achievement of Partial or Complete Remission of UPCR Through Week 12 and Through the End of Treatment
Description: Partial and complete remission were defined as follows:
  Partial remission (included all of the following):
  * Reduction from baseline by ≥50% in urine protein:creatinine ratio (UPCR)
  * Reduction in UPCR to a level that was <3.5 g/g
  * Subject could not have been a treatment failure
  Complete remission (included all of the following):
  * Reduction in UPCR to <0.3 g/g
  * Serum albumin within normal range
  * For subjects with abnormal serum creatinine levels at baseline, return to normal levels
  * For subjects with normal serum creatinine levels at baseline, final value within 20% of baseline levels
  * Subject could not have been a treatment failure
Time Frame: Baseline to week 12
Measure: Count of Participants; unit: Participants
Arm/Group | CCX140-B
Number analyzed (Participants) | 5
Participants
  No Complete or Partial remission at week 12/ end of treatment | 4
  Partial remission at Week 12 | 1

3. Secondary Outcome: Proportion of Subjects With Achievement of Complete Remission During the Treatment Period
Description: Complete remission is defined as reduction in urine protein:creatinine ratio (UPCR) to <0.3 g/g, normal serum albumin, and normal serum creatinine levels or within 20% of baseline levels.
Time Frame: Baseline to week 52
Measure: Count of Participants; unit: Participants
Arm/Group | CCX140-B
Number analyzed (Participants) | 5
Participants
  Achieved complete remission | 0
  Did not achieve complete remission | 5

4. Secondary Outcome: Time Taken of Subjects to Achieve Complete Remission During the Treatment Period
Description: as for outcome 3
Time Frame: Baseline to week 52
Measure: Number; unit: days
Arm/Group | CCX140-B
Number analyzed (Participants) | 5
days | NA — No subjects achieved complete remission

5. Secondary Outcome: Change From Baseline in Urine Protein:Creatinine Ratio (UPCR) Over Time
Description: Mean change from baseline in urinary protein:creatinine ratio (UPCR) over time.
Time Frame: Baseline to week 12 and week 52
Population: Data was not available for all patients at each timepoint
Measure: Mean (Standard Deviation); unit: g protein/g creatinine
Arm/Group | CCX140-B
Number analyzed (Participants) | 3
g protein/g creatinine
  Week 12 | -1.3100 (3.76247)
  Week 52: number analyzed (Participants) | 2
  Week 52 | -0.4985 (3.37926)

6. Secondary Outcome: Assessment of Time to and Proportion of Subjects With Achievement of Partial Remission During the Treatment Period
Description: Partial remission is defined as reduction from baseline by ≥50% in UPCR, reduction in UPCR to a level that was <3.5 g/g.
Time Frame: Baseline to week 52
Measure: Count of Participants; unit: Participants
Arm/Group | CCX140-B
Number analyzed (Participants) | 5
Participants
  Partial remission at Week 12 | 1
  Did not achieve partial remission | 4

7. Secondary Outcome: Time to Rescue Therapy
Description: Based on Investigator or physician initiation of glucocorticoids or new immunosuppressive agents or new major treatment modalities (e.g. plasmapheresis, dialysis)
Time Frame: Baseline to week 52
Population: Due to the small sample size and early termination of the study, no data could be collected
Arm/Group | CCX140-B
Number analyzed (Participants) | 0

8. Secondary Outcome: Mean Change From Baseline for eGFR Using the CKD-EPI Cystatin C Equation Over Time
Description: eGFR-Estimated Glomerular Filtration Rate;CKD-EPI=Chronic Kidney Disease Epidemiology Collaboration
Time Frame: Baseline to Week 12 and Week 52
Population: Data was not available for all patients at each timepoint
Measure: Mean (Full Range); unit: mL/min/1.73m²
Groups:
- CCX140-B: CCX140-B is an orally administered tablet. All enrolled subjects will initially be treated with the active study medication CCX140-B at a dose of 5 mg twice daily. Dose will increase in a step-wise fashion up to 15 mg twice daily.
Arm/Group | CCX140-B
Number analyzed (Participants) | 4
mL/min/1.73m²
  Week 12 | 7.50 [-11.0 to 37.0]
  Week 52: number analyzed (Participants) | 1
  Week 52 | -2.00 [-2.0 to -2.0]

9. Secondary Outcome: Mean Change From Baseline for the eGFR CKD-EPI Creatinine Equation Over Time
Description: CKD-EPI = Chronic Kidney Disease Epidemiology Collaboration; eGFR = estimated glomerular filtration rate
Time Frame: Baseline to Week 12 and Week 52
Population: Data was not available for all patients at each timepoint
Measure: Mean (Full Range); unit: ml/min/1.73 m²
Arm/Group | CCX140-B
Number analyzed (Participants) | 4
ml/min/1.73 m²
  Week 12 | -14.50 [-27.0 to -6.0]
  Week 52: number analyzed (Participants) | 1
  Week 52 | -15.0 [-15.0 to -15.0]

10. Secondary Outcome: Mean Change From Baseline for eGFR CKD-EPI Creatinine-Cystatin C Equation Over Time
Description: CKD-EPI = Chronic Kidney Disease Epidemiology Collaboration; eGFR = estimated glomerular filtration rate;
Time Frame: Baseline to Week 12 and Week 52
Population: Data was not available for all patients at each timepoint
Measure: Mean (Full Range); unit: ml/min/1.73 m²
Arm/Group | CCX140-B
Number analyzed (Participants) | 4
ml/min/1.73 m²
  Week 12 | -2.25 [-18.0 to 13.0]
  Week 52: number analyzed (Participants) | 1
  Week 52 | -8.0 [-8.0 to -8.0]

11. Secondary Outcome: Mean Change From Baseline for the MDRD Creatinine Equation Over Time
Description: MDRD = Modification of Diet in Renal Disease. The mean eGFR (using the MDRD Creatinine equation) change from baseline to Week 12 and Week 52
Time Frame: Baseline to Week 12 and Week 52
Population: Data was not available for all patients at each timepoint
Measure: Mean (Full Range); unit: ml/min/1.73 m²
Arm/Group | CCX140-B
Number analyzed (Participants) | 4
ml/min/1.73 m²
  Week 12 | -12.75 [-24.0 to -5.0]
  Week 52: number analyzed (Participants) | 1
  Week 52 | -13.00 [-13.00 to -13.00]

12. Secondary Outcome: Effect of CCX140-B Treatment on Quality of Life Endpoint SF-36V2
Description: Summary of the Effect of CCX140-B Treatment on Quality of Life Endpoints SF-36V2 for the overall trial
  SF-36v2: Medical Outcomes Survey Short Form-36 version 2.
  SF-36v2 measures each of the following eight health domains: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. Scores on each item are summed and averaged. The SF-36v2 component domain scores range from 0 (worst health) to 100 (best health).
Time Frame: Baseline to Week 52
Population: Due to the small sample size and early termination of the study, no data could be collected
Groups:
- CCX140-B: Drug: CCX140-B, orally administered tablet
Arm/Group | CCX140-B
Number analyzed (Participants) | 0

13. Secondary Outcome: Effect of CCX140-B Treatment on Quality of Life Endpoint EQ-5D-5L for the Overall Trial
Description: Summary of the Effect of CCX140-B Treatment on Quality of Life Endpoint EQ-5D-5L for the overall trial EQ-5D-5L: EuroQuality of Life-5 Domains-5 Levels. The EQ-5D-5L consists of : the EQ-5D descriptive system. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  The scale is numbered from 0 to 100. 100 means the best health you can imagine. 0 means the worst health you can imagine.
Time Frame: Baseline to Week 12 and Week 52
Population: Data was not available for all patients at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CCX140-B
Number analyzed (Participants) | 4
score on a scale
  Week 12 | 66.3 (31.98)
  Week 52: number analyzed (Participants) | 3
  Week 52 | 85 (0)

14. Secondary Outcome: Changes to Laboratory Parameters Related to Renal Function Including Serum Albumin, Creatinine, Cystatin C, Urinary Albumin:Creatinine Ratio, Total 24-hour Protein Excretion During the Trial
Description: Changes to laboratory parameters related to renal function including serum albumin, creatinine, cystatin C, urinary albumin:creatinine ratio, total 24-hour protein excretion during the trial
Time Frame: Baseline to Day 57
Population: No data collected
Arm/Group | CCX140-B
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | CCX140-B
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CCX140-B (N=5)
Amylase increased (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Blood potassium increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Fatigue (General disorders) | 1 (2)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (2)
Nasopharyngitis (Infections and infestations) | 1 (1)
Pulpitis dental (Infections and infestations) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Ophthalmoplegic migraine (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 1 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Tongue discomfort (Gastrointestinal disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
The CL012_140 study was terminated early due to lack of efficacy in another study, CL011_140, investigating the use of CCX140-B.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT03703908/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT03703908/SAP_001.pdf